CLINICAL TRIAL: NCT02099149
Title: Establishing a Sero-correlate of Protection Against Invasive Group B Streptococcus Disease in Newborns and Young Infants Aged Less Than 90 Days.
Brief Title: Antibody Levels Associated With Reduced Risk of Invasive Group B Streptococcus Disease in Infants Aged Less Than 90 Days
Status: Withdrawn | Type: Observational
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Other Study IDs: V98_28OB
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Invasive Group B Streptococcus Disease
Keywords: Group B Streptococcus; early onset disease; late onset disease; anticapsular antibodies; serotype specific
MeSH Terms: conditions — Late Onset Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Infants born to GBS colonized mother who do not develop GBS disease
- Cases: Infants with culture confirmed GBS disease

SUMMARY:
Compare anticapsular antibody levels against Group B Streptococcus at delivery in mothers and their infants who develop disease versus those who do not. Use this comparison to establish antibody levels associated with reductions in risk of GBS disease in infants aged less than 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending participating community/hospital antenatal clinics and/or delivering at participating delivery centers.
* Subjects aged ≥18 years.
* Able to understand and comply with planned study procedures.
* Provides written informed consent.

Exclusion Criteria:

* Refuses to consent to study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women aged 18 years or older attending for antenatal care or delivery at 3 academic hospital centers in the Johannesburg area and the antenatal clinics serving those hospital centers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Early onset Group B Streptococcus Disease due to serotypes Ia or III | 0-6 days
  Risk of early onset Group B Streptococcus disease (due to serotypes Ia or III) with respect to maternal or newborn anticapsular antibody levels at delivery

SECONDARY OUTCOMES:
Late onset Group B Streptococcus Disease due to serotype III | 7-90 days
  Risk of late onset Group B Streptococcus disease (due to serotypes III) with respect to maternal or newborn anticapsular antibody levels at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Respiratory and Meningeal Pathogen Research Unit, Soweto, Gauteng, South Africa